CLINICAL TRIAL: NCT04633642
Title: Cellular Proliferation, Dermal Repair, and Microbiological Effectiveness of Ultrasound Assisted Wound Debridement (UAW) Versus Standard Wound Treatment in Complicated Diabetic Foot Ulcers (DFU): A Randomized Controlled Trial
Brief Title: Ultrasound Assisted Wound Debridement (UAW) Versus Standard Wound Treatment in Complicated Diabetic Foot Ulcers (DFU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Francisco Javier Álvaro Afonso (Unknown); David Sevillano Fernández (Unknown); Yolanda García Álvarez (Unknown); Irene Sanz Corbalan (Unknown); Esther García Morales (Unknown)
Responsible Party: Principal Investigator, Jose Luis Lazaro Martinez, Prof.Dr, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.P. - C.I. 16/484-P
Record Dates: First submitted 2020-10-30; First posted 2020-11-18 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Diabetic Foot Ulcer
Keywords: ultrasound assisted wound debridement; surgical debridement; cellular proliferation; microbiology; diabetic foot ulcers
MeSH Terms: conditions — Diabetic Foot; Hyperplasia

STUDY DESIGN:
Intervention Model Description: A randomized and controlled parallel clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Group (UAW group) (Experimental): UAW debridement was performed using an UAW SONOCA 185 device (Söring GmbH, Germany). The UAW device generates an ultrasound low frequency of 25kHz and is equipped with three UAW instruments with different sonotrode shapes. The choice of sonotrode depends on wound depth, which ranges from superficial to deep. The UAW instrument piezoelectrically transforms the electrical energy delivered from the UAW device into mechanical oscillations in the sonotrode tip. For most wounds in the UAW group, a two-minute treatment with 40% intensity was performed by holding the sonotrode in contact mode, holding it perpendicular to the wound bed and moving it across in an up-and-down pattern.
  Interventions: Procedure: Ultrasound group
- Surgical group (Active Comparator): All debridement procedures were performed by the same surgeon (J.L.M.), who is specialist in diabetic foot surgery with more than 20 years of experience.
  Surgical debridement involved removal of all necrotic and devitalized tissue that was incompatible with healing, as well as surrounding callus.
  Interventions: Procedure: Surgical group

INTERVENTIONS:
Procedure: Ultrasound group — Every week during a six-week treatment period
  Arms: Ultrasound Group (UAW group)
Procedure: Surgical group — Every week during a six-week treatment period
  Arms: Surgical group

SUMMARY:
The investigators aimed to elucidate the effects of UAW debridement on cellular proliferation and dermal repair in complicated diabetic foot ulcers as compared to diabetic foot ulcers receiving surgical/sharp wound debridement. A randomized controlled trial was performed involving outpatients with complicated diabetic foot ulcers that either received surgical debridement or UAW debridement every week during a six-week treatment period.

DETAILED DESCRIPTION:
2. Methods

2.1. Trial design

A randomized and controlled parallel clinical trial was performed involving outpatients with complicated DFU that were admitted to specialized diabetic foot unit between November 2017 to December 2019. The study protocol received full approval from the Ethics Committee of the Hospital Clínico San Carlos, Madrid, Spain (C.P. - C.I. 16/484-P). Each patient provided written informed consent before inclusion.

2.1. Intervention

Participants were randomized and assigned to receive either surgical debridement or UAW debridement every week during a six-week treatment period.

Soft tissue punch biopsies (3mm) were taken after wound debridement sessions at week zero and week six.

2.2. Follow-up Patients were followed-up for 6 months after inclusion. During the follow-up period, the investigators recorded ulcer healing. Ulcer healing was defined as complete epithelialization without any sustained drainage up to 24 weeks after the end of the study follow-up.

2.3. Sample size The sample size was calculated using the Granmo v.12 program (Municipal Institute of Medical Research, Barcelona, Spain) (https://www.imim.cat/ofertadeserveis/software-public/granmo/ ). Therefore, we analyzed 51 patients (24 in surgical group and 27 en UAW group) with an alpha of 0.05 and a statistical power of 0.80.

2.4. Randomization A computer-generated random number table was used to carry out the randomization of the patients into the two groups by an investigator who was blinded to the identity of the participants.

2.5. Blinding None of the participants, care providers, and outcome adjudicators was blinded to the interventions after assignment.

2.6. Statistical Analysis Statistical analysis was performed using SPSS for IOs version 21.0 (SPSS, Inc. Chicago, IL, USA). The assumption of normality of all continuous variables was verified using the Kolmogorov-Smirnov test. Statistical differences between groups were calculated using the Chi-Square test and, where appropriate, Fisher's exact test for categorical variables. The Mann-Whitney U test was performed for abnormally distributed quantitative parameters, and Student's t-test was performed for quantitative variables that were distributed normally. The criteria of p < 0.05 was accepted as statistically significant with a confidence interval of 95%.

This study was conducted in accordance with the Declaration of Helsinki (2013 revision) and followed all local laws and regulations in clinical research investigations in patients.

ELIGIBILITY:
Inclusion Criteria:

* • Male and female patients ≥18 years old

  * Type 1 or type 2 diabetes with levels of HbA1c≤85.8 mmol/mol (10%) within 30 days of the beginning of the study
  * Wound stages IB, IIB, ID, and IID according to the University of Texas Diabetic Wound Classification [11]
  * Wound duration of 1-24 months
  * Wound size between 1-30 cm2 after debridement
  * Clinical picture of wounds showing mild or moderate infection, according to the criteria of the Infectious Disease Society of America Guidelines [12] and the European Wound Management Association (EWMA) [13]
  * Ankle-brachial index (ABI) ≤0.9 and ankle systolic blood pressure (ASBP) ≥70mmHg, or toe systolic blood pressure (TSBP) ≥50mmHg, ABI>0.9, TSBP ≥50mmHg and toe-brachial index (TBI) ≤0.7

Exclusion Criteria:

* • Chronic renal disease or dialysis

  * Non-treated osteomyelitis
  * Necrotizing soft tissue infections
  * Critical limb ischaemia patients with ABI≤0.5 and ASBP<70mmHg or <50mmHg
  * Life expectancy <6 months due to malignant DFU
  * Pregnancy and lactation
  * Patients diagnosed with hepatitis or human immunodeficiency virus (HIV)
  * Patients showing local or systemic conditions that may impair tissue repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lázaro Martinez, Professor, Principal Investigator — Universidad Complutense de Madrid
Locations (2):
- Spain (2):
  - Fancisco Javier Álvaro Afonso, Madrid
  - José Luis Lázaro Martínez, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schaper NC, van Netten JJ, Apelqvist J, Bus SA, Hinchliffe RJ, Lipsky BA; IWGDF Editorial Board. Practical Guidelines on the prevention and management of diabetic foot disease (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3266. doi: 10.1002/dmrr.3266. PMID 32176447
- [Background] Kim PJ, Steinberg JS. Wound care: biofilm and its impact on the latest treatment modalities for ulcerations of the diabetic foot. Semin Vasc Surg. 2012 Jun;25(2):70-4. doi: 10.1053/j.semvascsurg.2012.04.008. PMID 22817855
- [Background] Kingsley A, Lewis T, White R. Debridement and wound biofilms. J Wound Care. 2011 Jun;20(6):286. No abstract available. PMID 21739682
- [Background] Swanson T, Lazaro-Martinez JL, Braumann C, Kirchhoff JB, Gachter B, van Acker K. Ultrasonic-assisted wound debridement: report from a closed panel meeting. J Wound Care. 2020 Feb 2;29(2):128-135. doi: 10.12968/jowc.2020.29.2.128. PMID 32058848
- [Background] Rayman G, Vas P, Dhatariya K, Driver V, Hartemann A, Londahl M, Piaggesi A, Apelqvist J, Attinger C, Game F; International Working Group on the Diabetic Foot (IWGDF). Guidelines on use of interventions to enhance healing of chronic foot ulcers in diabetes (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3283. doi: 10.1002/dmrr.3283. PMID 32176450
- [Background] Lazaro-Martinez JL, Alvaro-Afonso FJ, Garcia-Alvarez Y, Molines-Barroso RJ, Garcia-Morales E, Sevillano-Fernandez D. Ultrasound-assisted debridement of neuroischaemic diabetic foot ulcers, clinical and microbiological effects: a case series. J Wound Care. 2018 May 2;27(5):278-286. doi: 10.12968/jowc.2018.27.5.278. PMID 29738301
- [Background] Altland OD, Dalecki D, Suchkova VN, Francis CW. Low-intensity ultrasound increases endothelial cell nitric oxide synthase activity and nitric oxide synthesis. J Thromb Haemost. 2004 Apr;2(4):637-43. doi: 10.1111/j.1538-7836.2004.00655.x. PMID 15102020
- [Background] Driver VR, Yao M. Discussion. Current status of the use of modalities in wound care: electrical stimulation and ultrasound therapy. Plast Reconstr Surg. 2011 Jan;127 Suppl 1:103S-104S. doi: 10.1097/PRS.0b013e3182050c35. No abstract available. PMID 21200279
- [Background] Ennis WJ, Foremann P, Mozen N, Massey J, Conner-Kerr T, Meneses P. Ultrasound therapy for recalcitrant diabetic foot ulcers: results of a randomized, double-blind, controlled, multicenter study. Ostomy Wound Manage. 2005 Aug;51(8):24-39. PMID 16234574
- [Background] Driver VR, Yao M, Miller CJ. Noncontact low-frequency ultrasound therapy in the treatment of chronic wounds: a meta-analysis. Wound Repair Regen. 2011 Jul-Aug;19(4):475-80. doi: 10.1111/j.1524-475X.2011.00701.x. Epub 2011 Jun 7. PMID 21649783
- [Background] Armstrong DG, Lavery LA, Harkless LB. Validation of a diabetic wound classification system. The contribution of depth, infection, and ischemia to risk of amputation. Diabetes Care. 1998 May;21(5):855-9. doi: 10.2337/diacare.21.5.855. PMID 9589255
- [Background] Lipsky BA, Berendt AR, Cornia PB, Pile JC, Peters EJ, Armstrong DG, Deery HG, Embil JM, Joseph WS, Karchmer AW, Pinzur MS, Senneville E; Infectious Diseases Society of America. 2012 Infectious Diseases Society of America clinical practice guideline for the diagnosis and treatment of diabetic foot infections. Clin Infect Dis. 2012 Jun;54(12):e132-73. doi: 10.1093/cid/cis346. PMID 22619242
- [Background] Boulton AJ, Armstrong DG, Albert SF, Frykberg RG, Hellman R, Kirkman MS, Lavery LA, Lemaster JW, Mills JL Sr, Mueller MJ, Sheehan P, Wukich DK; American Diabetes Association; American Association of Clinical Endocrinologists. Comprehensive foot examination and risk assessment: a report of the task force of the foot care interest group of the American Diabetes Association, with endorsement by the American Association of Clinical Endocrinologists. Diabetes Care. 2008 Aug;31(8):1679-85. doi: 10.2337/dc08-9021. No abstract available. PMID 18663232
- [Background] Tan T, Shaw EJ, Siddiqui F, Kandaswamy P, Barry PW, Baker M; Guideline Development Group. Inpatient management of diabetic foot problems: summary of NICE guidance. BMJ. 2011 Mar 23;342:d1280. doi: 10.1136/bmj.d1280. No abstract available. PMID 21430002
- [Background] Bus SA, Armstrong DG, Gooday C, Jarl G, Caravaggi C, Viswanathan V, Lazzarini PA; International Working Group on the Diabetic Foot (IWGDF). Guidelines on offloading foot ulcers in persons with diabetes (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3274. doi: 10.1002/dmrr.3274. PMID 32176441
- [Background] Tardaguila-Garcia A, Lazaro-Martinez JL, Sanz-Corbalan I, Garcia-Alvarez Y, Alvaro-Afonso FJ, Garcia-Morales E. Correlation between Empirical Antibiotic Therapy and Bone Culture Results in Patients with Osteomyelitis. Adv Skin Wound Care. 2019 Jan;32(1):41-44. doi: 10.1097/01.ASW.0000542527.48815.1f. PMID 30376455
- [Background] Wang D, Stockard CR, Harkins L, Lott P, Salih C, Yuan K, Buchsbaum D, Hashim A, Zayzafoon M, Hardy RW, Hameed O, Grizzle W, Siegal GP. Immunohistochemistry in the evaluation of neovascularization in tumor xenografts. Biotech Histochem. 2008 Jun;83(3-4):179-89. doi: 10.1080/10520290802451085. PMID 18846440
- [Background] Achar RA, Silva TC, Achar E, Martines RB, Machado JL. Use of insulin-like growth factor in the healing of open wounds in diabetic and non-diabetic rats. Acta Cir Bras. 2014 Feb;29(2):125-31. doi: 10.1590/S0102-86502014000200009. PMID 24604317
- [Background] Wollina U, Schmidt WD, Kronert C, Nelskamp C, Scheibe A, Fassler D. Some effects of a topical collagen-based matrix on the microcirculation and wound healing in patients with chronic venous leg ulcers: preliminary observations. Int J Low Extrem Wounds. 2005 Dec;4(4):214-24. doi: 10.1177/1534734605283001. PMID 16286373
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Maan ZN, Januszyk M, Rennert RC, Duscher D, Rodrigues M, Fujiwara T, Ho N, Whitmore A, Hu MS, Longaker MT, Gurtner GC. Noncontact, low-frequency ultrasound therapy enhances neovascularization and wound healing in diabetic mice. Plast Reconstr Surg. 2014 Sep;134(3):402e-411e. doi: 10.1097/PRS.0000000000000467. PMID 25158717
- [Background] Roper JA, Williamson RC, Bally B, Cowell CAM, Brooks R, Stephens P, Harrison AJ, Bass MD. Ultrasonic Stimulation of Mouse Skin Reverses the Healing Delays in Diabetes and Aging by Activation of Rac1. J Invest Dermatol. 2015 Nov;135(11):2842-2851. doi: 10.1038/jid.2015.224. Epub 2015 Jun 16. PMID 26079528
- [Background] Butcher G, Pinnuck L. Wound bed preparation: ultrasonic-assisted debridement. Br J Nurs. 2013 Mar 28-Apr 10;22(6):S36, S38-43. doi: 10.12968/bjon.2013.22.Sup4.S36. PMID 23587975
- [Background] Michailidis L, Bergin SM, Haines TP, Williams CM. A Systematic Review to Compare the Effect of Low-frequency Ultrasonic Versus Nonsurgical Sharp Debridement on the Healing Rate of Chronic Diabetes-related Foot Ulcers. Ostomy Wound Manage. 2018 Sep;64(9):39-46. PMID 30256750
- [Background] Michailidis L, Bergin SM, Haines TP, Williams CM. Healing rates in diabetes-related foot ulcers using low frequency ultrasonic debridement versus non-surgical sharps debridement: a randomised controlled trial. BMC Res Notes. 2018 Oct 16;11(1):732. doi: 10.1186/s13104-018-3841-4. PMID 30326972
- [Background] Messa CA 4th, Chatman BC, Rhemtulla IA, Broach RB, Mauch JT, D'Angelantonio AM 3rd, Fischer JP. Ultrasonic debridement management of lower extremity wounds: retrospective analysis of clinical outcomes and cost. J Wound Care. 2019 May 1;28(Sup5):S30-S40. doi: 10.12968/jowc.2019.28.Sup5.S30. PMID 31067172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label randomized and controlled parallel clinical trial was performed involving outpatients with complicated Diabetic Foot Ulcer that were admitted to specialized diabetic foot unit between November 2017 to December 2019.
Pre-assignment Details: 51 patients met inclusion criteria and were were randomized to treatment
Groups:
- Ultrasound Group (UAW Group): For most wounds in the UAW group, a two-minute treatment with 40% intensity was performed by holding the sonotrode in contact mode, holding it perpendicular to the wound bed and moving it across in an up-and-down pattern. Every week during 6 weeks
- Surgical Group: Surgical debridement involved removal of all necrotic and devitalized tissue that was incompatible with healing, as well as surrounding callus. Every week during 6 weeks
Period: Overall Study
Arm/Group | Ultrasound Group (UAW Group) | Surgical Group
Started (November 2017) | 27 (27 participants) | 24 (24 participants)
Completed (December 2019) | 26 (26 participants) | 22 (22 participants)
Not Completed | 1 | 2
Not completed — Chronic renal disease, critical limb ischemia and heart attack | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Ultrasound Group (UAW Group): UAW debridement was performed using an UAW SONOCA 185 device (Söring GmbH, Germany). The UAW device generates an ultrasound low frequency of 25kHz and is equipped with three UAW instruments with different sonotrode shapes. The choice of sonotrode depends on wound depth, which ranges from superficial to deep. The UAW instrument piezoelectrically transforms the electrical energy delivered from the UAW device into mechanical oscillations in the sonotrode tip. For most wounds in the UAW group, a two-minute treatment with 40% intensity was performed by holding the sonotrode in contact mode, holding it perpendicular to the wound bed and moving it across in an up-and-down pattern.
  Ultrasound group: For most wounds in the UAW group, a two-minute treatment with 40% intensity was performed by holding the sonotrode in contact mode, holding it perpendicular to the wound bed and moving it across in an up-and-down pattern. For wounds measuring >15cm2, the debridement procedure was increased to three minutes. In addition to UAW debridement, a scalpel was used for careful tissue removal, but only if periwound skin exhibited calluses and maceration.
- Surgical Group: All debridement procedures were performed by the same surgeon (J.L.M.), who is specialist in diabetic foot surgery with more than 20 years of experience.
  Surgical debridement involved removal of all necrotic and devitalized tissue that was incompatible with healing, as well as surrounding callus.
  Ultrasound group: For most wounds in the UAW group, a two-minute treatment with 40% intensity was performed by holding the sonotrode in contact mode, holding it perpendicular to the wound bed and moving it across in an up-and-down pattern. For wounds measuring >15cm2, the debridement procedure was increased to three minutes. In addition to UAW debridement, a scalpel was used for careful tissue removal, but only if periwound skin exhibited calluses and maceration.
- Total: Total of all reporting groups
Arm/Group | Ultrasound Group (UAW Group) | Surgical Group | Total
Number analyzed (Participants) | 27 | 24 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 22 | 46
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (12.4) | 58 (5.4) | 61.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 24 | 24 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 24 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — 51 outpatients with complicated diabetic foot ulcer were admitted to specialized diabetic foot unit in Spain
  participants
    Spain | 27 | 24 | 51
Type Diabetes Mellitus [Count of Participants; unit: Participants]
  Type 1 | 5 | 0 | 5
  Type 2 | 22 | 24 | 46
Duration of Diabetes [Mean (Standard Deviation); unit: years] — Duration of diabetes in years
  years | 22 (12.9) | 10.3 (5.0) | 16.15 (8.95)
Glycated hemoglobin [Mean (Standard Deviation); unit: mmol/L] — Glycated hemoglobin in mmol/L
  mmol/L | 57 (9.9) | 51 (4.5) | 54 (9.4)
Texas Classification [Count of Participants; unit: Participants] — The University of Texas system for ulcer classification primarily grades ulcers based on depth; each grade is then 'staged', which divides patients who have infected ulcers, those who have ischaemia and those who have both infection and ischaemia.
  IB: Superficial wound with infection. IIB: Deep wound with infection. ID: Superficial wound with infection and ischaemia. IID: Deep wound with infection and ischaemia.
  Grades IIB and IID were considered worse outcomes
  Participants
    IB | 4 | 4 | 8
    II B | 3 | 8 | 11
    ID | 12 | 8 | 20
    IID | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Neo-angiogenesis (Microvessel Density) at 6 Weeks
Description: Sections of tissue were immunohistochemically-stained with the CD31 marker. Light microscopy was used to count the number of microvessels/endothelial cells in a standardized grid, with the results expressed as microvessel density (Leica DMD 800 morphometric system). Microvessel density was scored according to the following scale: 0 (absent), 1 (low, at least one microvessel), 2 (moderate) and 3 (more than two micro vessels).
  Higher scores mean a better outcome
Time Frame: At week zero and week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultrasound Group (UAW Group) | Surgical Group
Number analyzed (Participants) | 27 | 24
score on a scale | 2.82 (0.52) | 1.77 (1.30)
Statistical Analysis 1: Comparison: Ultrasound Group (UAW Group) vs Surgical Group; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney) — The threshold for statistical significances was p<0.05; Mean Difference (Final Values) = 1.05, Standard Deviation 0.74

2. Primary Outcome: Change From Baseline Collagen Formation (Collagen Content ) at 6 Weeks
Description: Massons's trichome staining was used to differentiate collagen content from other components, such as muscle fibrin and erythrocytes, in tissue samples. Collagen content was scored according to the following scale: 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Higher scores mean a better outcome.
Time Frame: At week zero and week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultrasound Group (UAW Group) | Surgical Group
Number analyzed (Participants) | 27 | 24
score on a scale | 2.81 (0.48) | 1.20 (0.26)
Statistical Analysis 1: Comparison: Ultrasound Group (UAW Group) vs Surgical Group; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p<0.05; Mean Difference (Final Values) = 1.61, Standard Deviation 0.17

3. Primary Outcome: Change From Baseline Myofibroblasts Formation (Myofibroblasts Content) at 6 Weeks
Description: Actin staining was used to evaluate the presence of myofibroblasts involved in wound healing. These cells increase in number during wound healing. The number of stained cells was semi-quantitatively analyzed using a 0 - 3 scaling score (0= no myofibroblasts, 1= myofibroblasts in low quantity, 2= myofibroblasts in moderate quantity, 3= myofibroblasts in high quantity)
Time Frame: At week zero and week 6
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ultrasound Group (UAW Group) | Surgical Group
Number analyzed (Participants) | 27 | 24
score on a scale | 2.56 (0.89) | 2.00 (0.10)
Statistical Analysis 1: Comparison: Ultrasound Group (UAW Group) vs Surgical Group; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.56, Standard Deviation 0.79

4. Secondary Outcome: Comparison of Quantitative Microbiological Analysis (Bacterial Counts Expressed Colony-forming Units Per Gram of Tissue) (CFU/g)
Description: Tissue samples were weighed and mechanically homogenised in 0.5ml volumes of sterile phosphate buffered saline (PBS, Sigma Aldrich, St Louis, MO). Homogenates were diluted and plated onto Columbia agar (BD, Sparks, MD), Columbia agar supplemented with colistin and nalidixic acid (BD), MacConkey agar (BD), and Sabouraud dextrose agar (BD) using a spiral plater workstation (Don Whitley Scientific, Shipley, UK).The limit of detection was 10 colony-forming units (CFU). Results were expressed as CFU per gram of tissue (CFU/g). Isolated microorganisms were identified by standard criteria and the BBL Crystal identification system (BD). Susceptibility testing of Staphylococcus aureus isolates for oxacillin was performed according to Clinical and Laboratory Standards Institute (CLSI) guidelines, using a 30g cefoxitin disc and Mueller-Hinton agar .
Time Frame: At week zero and week 6
Measure: Mean (Standard Deviation); unit: Log10 CFU/g
Arm/Group | Ultrasound Group (UAW Group) | Surgical Group
Number analyzed (Participants) | 27 | 24
Log10 CFU/g | 2.11 (0.8) | 4.39 (1.24)
Statistical Analysis 1: Comparison: Ultrasound Group (UAW Group) vs Surgical Group; We analyzed 51 patients (24 in surgical group and 27 in UAW group) with a statistical power of 0.80 and an alpha of 0.05, with a power of the clinical di↵erence of 37% to detect a statistically significant between groups; Test type: Superiority; p = 0.01, t-test, 2 sided — The threshold for statistical significance was p<0.05; Mean Difference (Final Values) = -2.28, Standard Deviation 0.44

5. Secondary Outcome: Wound Score at 6 Weeks
Description: Wound bed tissue was evaluated for presence, quality, and consistency of granulation tissue using a validated wound scoring system, with scores ranging between a minimum of zero points and maximum of seven points. Higher scores mean a better outcome.
Time Frame: Six weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultrasound Group (UAW Group) | Surgical Group
Number analyzed (Participants) | 27 | 24
score on a scale | 5.4 (1.5) | 5.6 (0.7)
Statistical Analysis 1: Comparison: Ultrasound Group (UAW Group) vs Surgical Group; Test type: Superiority; p = 0.93, t-test, 2 sided — The threshold for statistics significance was p<0.05; Mean Difference (Final Values) = 0.2

6. Secondary Outcome: Wound Size
Description: A planimetric measurements of wound size were conducted using Visitrak (Smith & Nephew, Hull, UK), with the area of the lesion determined with an approximation of ±5mm2
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Centimeter square
Arm/Group | Ultrasound Group (UAW Group) | Surgical Group
Number analyzed (Participants) | 27 | 24
Centimeter square | 1.0 (1.22) | 0.88 (1.04)
Statistical Analysis 1: Comparison: Ultrasound Group (UAW Group) vs Surgical Group; We analyzed 51 patients (24 in surgical group and 27 in UAW group) with a statistical power of 0.80 and an alpha of 0.05, with a power of the clinical difference of 37% to detect a statistically significant between groups; Test type: Superiority; p = 0.711, t-test, 2 sided; Mean Difference (Final Values) = 0.02, Standard Deviation 0.18

ADVERSE EVENTS:
Time Frame: 6 months after inclusion
Arm/Group | Ultrasound Group (UAW Group) | Surgical Group
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/24
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24
Other Adverse Events (participants affected / at risk) | 0/27 | 0/24

LIMITATIONS AND CAVEATS:
Future trials may also evaluate efficiency or cost-effectiveness of both treatments

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04633642/Prot_SAP_000.pdf